CLINICAL TRIAL: NCT06634576
Title: Assessing the Reliability of Smooth Pursuit Across Various Neck Postures Using a Custom Ocular Motor Detection System
Acronym: Ocular motor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Jeng-Heng Lin, Principal Investigator, Kaohsiung Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KMUHIRB-F(II)-20210114
Record Dates: First submitted 2024-09-22; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Ocular Motor Detectation; Vestibular; Cervicogenic Dizziness; Oculomotor System
Keywords: Oculomotor system; Vestibular; cervicogenic dizziness; Ocular motor detectation

STUDY DESIGN:
Intervention Model Description: All for health populations.
  Inclusion criterias following:
  1. Age between 20 and 60 years.
  2. No history of significant neck surgeries.
  3. No history of corrective eye surgery.
  4. No skeletal muscle injuries or pain in the upper or lower limbs.
  5. Free from vestibular system-related disorders and neurological symptoms.
  6. Participants must avoid food and drink for 3 hours before the experiment.
  7. Participants should have 8 hours of sleep the night before the experiment.
  Exclusion criterias following:
  1. Any participant who has undergone vision correction surgery in the last year.
  2. Any participant who has experienced significant head or neck trauma in the past year.
  3. Any participant with a history of vestibular system disorders or neurological symptoms.
  4. Participants who have used medications or alcohol for an extended period.
  5. Participants with abnormal pain in any part of the torso.
  6. Individuals suffering from claustrophobia.
Masking Description: In research protocol, all neck postures were randomized, and did eye tracker recalibration before each task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health population (Experimental): Used custom-made ocular motor system to adjust the neck postures of participants, to examine the reliability of data and compared the pursuit ability in three different neck motion planes, seven different neck postures.
  Interventions: Device: Smooth pursuit neck torsion test

INTERVENTIONS:
Device: Smooth pursuit neck torsion test — Used custom-made system to stimulate the procedure of smooth pursuit neck torsion test in the current study, the multiple axis motion platform can adjust the neck postures to three different neck motion planes, seven different neck postures.

SUMMARY:
Background and Purpose: The assessment of ocular motor control through the manipulation of diverse sensory stimuli can facilitate the diagnosis of dizziness. However, the testing process typically encompasses a single rotational axis. This study aims to investigate the performance of ocular motor control under multi-axis neck rotation postures. To verify the data quality performance and reliability of the custom-made ocular motor features detection system, validate the consistency of system eye movement parameters, and investigate the effect of different neck plane positions on tracking performance. Methods: A total of seven healthy volunteers participated in this study. The study involved ocular motor tracking tasks in different neck positions with all seven subjects, A total of seven subjects were examined, comprising neutral neck posture, left lateral flexion posture, right lateral flexion posture, neck extension posture, neck flexion posture, left neck torsion posture, and right neck torsion posture. The study evaluated eye movement parameters in different planes, including Gain (representing pursuit speed), SPNTD (representing pursuit differences across planes), Accuracy (representing pursuit accuracy), and Latency (representing pursuit latency), as well as the reliability of these parameters. The reliability of the parameters was verified using the intraclass coefficient (ICC). Non-parametric tests (Friedman test) were used to verify the performance of ocular motor tracking in different neck positions, and post-hoc analysis (Wilcoxon sign test) was used to verify statistical differences.

DETAILED DESCRIPTION:
The assessment of ocular motor control through the manipulation of various sensory stimuli helps diagnose dizziness. However, most existing tests focus solely on a single rotational axis. This study aims to evaluate the performance of ocular motor control under multi-axis neck rotation postures. The research objective was integrated the desktop eye tracker with a six-axis Stewart platform to establish an ocular motor features detection system. This system will be used to validate the consistency of the system in ocular motor parameters and explore how different neck plane positions affect tracking performance.

Methods:

The smooth pursuit task was conducted under seven different neck postures:

1. Neutral neck posture
2. Left lateral flexion posture 3, Right lateral flexion posture 4, Neck extension posture

5. Neck flexion posture 6. Left neck torsion posture 7. Right neck torsion posture For each posture, participants were seated in a chair with their heads fixed in position to prevent any movement that could stimulate the vestibular system. The Stewart platform was used to control the neck posture of the participant by moving their body, allowing for specific neck rotations or flexions without moving the head. This setup ensured the focus remained solely on the effect of neck posture on smooth pursuit eye movements.

Participants were asked to track a light point moving horizontally across the screen in a sinusoidal trajectory. The target's movement was designed based on Simple Harmonic Motion (SHM) to allow for smooth, continuous movement that minimizes abrupt stops, which can trigger saccadic eye movements (quick, jerky movements). SHM was chosen because it better matches the natural movement of smooth pursuit eye tracking.

The target speed was set at 30° per second, and the amplitude of the target's movement ranged from 30° to 40°, based on previous studies indicating that these values were optimal for distinguishing between healthy individuals and those with vestibular or cervical dysfunction. The task required participants to follow the moving target as closely and smoothly as possible, while their eye movements were recorded using the Gaze-point 3 (GP3) eye tracker, which sampled at 60Hz.

Key Parameters Recorded:

1. Gain: This parameter represents the ratio of eye velocity to target velocity, effectively measuring how well the eyes can match the speed of the moving target. A gain of 1 indicates perfect pursuit, while values less than 1 indicate that the eyes are lagging behind the target.
2. SPNTD: This parameter (Smooth Pursuit Neck Torsion Difference) compares the smooth pursuit performance in neutral neck posture to that in various torsional neck postures. It helps to evaluate the impact of different neck positions on smooth pursuit abilities.
3. Accuracy: This measures how precisely the eyes follow the target. It reflects the angular error between the actual eye position and the position of the moving target at any given time.
4. Latency: This parameter measures the delay in the onset of smooth pursuit after the target begins moving. A lower latency indicates a faster response, which is important for evaluating the ability of participants to start tracking the target quickly and smoothly.

Data Analysis:

The reliability of the system and the parameters mentioned above were evaluated using the Intraclass Correlation Coefficient (ICC). The ICC was calculated for gain, SPNTD, accuracy, and latency to assess how consistently the participants; smooth pursuit performance could be measured across different neck postures.

Additionally, a Friedman test (a non-parametric test) was conducted to determine whether there were statistically significant differences in smooth pursuit performance across the various neck postures. For positions that showed significant differences, Wilcoxon signed-rank tests (a post-hoc analysis) were applied to identify which specific neck postures resulted in significant changes in smooth pursuit performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 60 years.
2. No history of significant neck surgeries.
3. No history of corrective eye surgery.
4. No skeletal muscle injuries or pain in the upper or lower limbs.
5. Free from vestibular system-related disorders and neurological symptoms.
6. Participants must avoid food and drink for 3 hours before the experiment.
7. Participants should have 8 hours of sleep the night before the experiment.

Exclusion Criteria:

1. Any participant who has undergone vision correction surgery in the last year.
2. Any participant who has experienced significant head or neck trauma in the past year.
3. Any participant with a history of vestibular system disorders or neurological symptoms.
4. Participants who have used medications or alcohol for an extended period.
5. Participants with abnormal pain in any part of the torso.
6. Individuals suffering from claustrophobia.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Analyzied the reliability of custom-made ocular motor detectation system | From enrollment to the end of research at 1 day.
  The custom-made system would output four parameters in this study. Used Intraclass correlation coefficient (ICC) to examine the reliability of pursuit parameters.

SECONDARY OUTCOMES:
Examine the pursuit ability in seven different neck postures. | From enrollment to the end of treatment at 1 day
  A custom-made system would change the neck posture in seven different neck postures. Used nonparametric(Friedman test) to analyze the pursuit ability in seven different neck postures, if the results were significant(p-value less than 0.05), used Wilcoxon sign rank to be the posthoc test.

CONTACTS AND LOCATIONS:
Overall Officials: Guo Lan-Yuen Guo, Lan-Yuen, Professor, Phd, Study Chair — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Sanmin District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual information(e.g age, born, research date) Personal pursuit ability results in the current study, like pursuit synchronized in each neck posture, the difference of pursuit synchronized in each neck motion plane, pursuit accuracy, potential pursuit reaction time.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 3 years after the publication of results.